CLINICAL TRIAL: NCT04824599
Title: Interpectoral and Pectoserratus Plane Block vs Local Anesthetic Infiltration for Partial Mastectomy - a Prospective Randomized Trial
Brief Title: Regional Anesthesia and Partial Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Patryk Eisler, Consultant in Anesthesiology and Intensive care, Karlstad Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIVFOU-930411
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasm
Keywords: Segmental Mastectomy,; Analgesia; Regional anesthesia; Breast surgery
MeSH Terms: conditions — Breast Neoplasms; Agnosia | interventions — Ropivacaine; Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS+subcutaneus local anesthetic infiltration (Active Comparator): Preoperative ultrasound-led PECS II blockade with ropivacaine 3,75mg/ml (2mg/kg). After surgery - wound infiltration by the surgeon with ropivacaine 2mg/ml (1mg/kg).
  Interventions: Procedure: PECS II; Procedure: Subcutaneus local anesthetic infiltration; Drug: Ropivacaine; Device: bk medical Flex Focus 500 Ultrasound Machine
- Local anesthetic infiltration (Active Comparator): Prior to scrubbing surgeon infiltrates the thought incision area with ropivacaine 3,75/ml (1mg/kg). Perioperatively after removal of the tumor follows the deep infiltration of the wound with ropivacaine 3,75mg/ml (2mg/kg).
  Interventions: Procedure: Local anesthetic infiltration; Drug: Ropivacaine

INTERVENTIONS:
Procedure: PECS II — Pectoral nerves block (PECS II) is performed with the help of ultrasound. Two injection are performed in two fascial planes. One between pectoralis major muscle and serratus anterior muscle. Second one between pectoralis major and minor muscles.
  Other Names: Pectoral nerves block
  Arms: PECS+subcutaneus local anesthetic infiltration
Procedure: Local anesthetic infiltration — Ropivacaine is administered by surgeon prior to scrubbing and following the removal of the tumor.
  Arms: Local anesthetic infiltration
Procedure: Subcutaneus local anesthetic infiltration — Ropivacaine is administered by the surgeon at the end of surgery
  Arms: PECS+subcutaneus local anesthetic infiltration
Drug: Ropivacaine — Local anesthetic ropivacaine is administered in both study arms according to the study protocol
  Other Names: Local anesthetic
Device: bk medical Flex Focus 500 Ultrasound Machine — Ultrasound with linear probe is performed. Using in-plane technique a correct placement of the injection needle is secured.
  Other Names: High Frequency Linear 8870 probe
  Arms: PECS+subcutaneus local anesthetic infiltration

SUMMARY:
Pectoralis nerves plane block (PECS) first described by Blanco in 2011 has become part of postoperative pain management in breast surgery, thoracic surgery and thoracic trauma. The combination of low complication risk and easiness in mastering of PECS block has made it an interesting alternative to thoracic epidural anesthesia (TEDA) and paravertebral blockade (PVB) for pain treatment after breast surgery. Several studies showed good results when PECS was compared to PVB. PECS blockade however is a procedure requiring some resources in the operating room. An alternative approach is to inject local anesthetics (LA) in the operation field by the surgeon.

The hypothesis' tested in this study is primarily: that PECS blockade is superior to LA being injected by surgeon in the operating field measured by end points such as: post-operative pain, post-operative analgesics use, post-operative nausea or vomiting (PONV) and length of stay in the post anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for partial mastectomy (lumpectomy).

Exclusion Criteria:

* Scheduled cryosection
* Axillary node dissection
* Re-resection
* Age under 18 or unable to give an informed concent
* Chronic pain history
* Allergy to local anesthetics
* History of active drug addiction
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
maximal pain in PACU measured with 11 point numerical rating scale (NRS) | measured at discharge from PACU (on average 4 hours).
  NRS scale is a validated for assessment of pain. It is a 11 point scale (0-10) used to estimate severity of postoperative pain. On NRS scale the higher value indicates more severe symptoms.
Intraoperative fentanyl use | Time is measured from start of the anesthesia until discharge to PACU (on average 3 hours)
  dose of fentanyl used during surgery in milligrams [mg].

SECONDARY OUTCOMES:
Postoperative analgesic use | measured at 24 hours postoperatively.
  Postoperative analgesic use is related to pain severity and can be a factor leading to increased length of stay in PACU.
Maximal postoperative nausea and vomiting(PONV) in PACU measured with 11 point numerical rating scale (NRS) | measured at discharge from PACU (on average 4 hours).
  PONV NRS similar to pain NRS is an 11 point scale (0-10) used to estimate severity of postoperative nausea. On NRS scale the higher value indicates more severe symptoms.
Length of stay in PACU | on average 4 hours.
  Is an dependant of multiple factors and an important measurement that can indicate beneficial therapeutic choice.
Maximal postoperative nausea and vomiting(PONV) after discharge from PACU measured with 11 point numerical rating scale (NRS) | 24 hours
  PONV NRS similar to pain NRS is an 11 point scale used to estimate severity of postoperative nausea.
Maximal pain after discharge from PACU measured with 11 point numerical rating scale (NRS) | 24 hours
  NRS scale is a validated for assessment of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ragnar Henningsson, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Central Hospital in Karlstad, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs A, Lemoine A, Joshi GP, Van de Velde M, Bonnet F; PROSPECT Working Group collaborators#. PROSPECT guideline for oncological breast surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2020 May;75(5):664-673. doi: 10.1111/anae.14964. Epub 2020 Jan 26. PMID 31984479
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Apfel CC, Roewer N, Korttila K. How to study postoperative nausea and vomiting. Acta Anaesthesiol Scand. 2002 Sep;46(8):921-8. doi: 10.1034/j.1399-6576.2002.460801.x. PMID 12190791
- [Background] Woodworth GE, Ivie RMJ, Nelson SM, Walker CM, Maniker RB. Perioperative Breast Analgesia: A Qualitative Review of Anatomy and Regional Techniques. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):609-631. doi: 10.1097/AAP.0000000000000641. PMID 28820803
- [Background] Habib AS, Kertai MD, Cooter M, Greenup RA, Hwang S. Risk factors for severe acute pain and persistent pain after surgery for breast cancer: a prospective observational study. Reg Anesth Pain Med. 2019 Feb;44(2):192-199. doi: 10.1136/rapm-2018-000040. Epub 2019 Jan 5. PMID 30700614
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Derived] Eisler P, Zimmermann S, Henningsson R. Interpectoral and Pectoserratus Plane Block vs. Local Anesthetic Infiltration for Partial Mastectomy: A Prospective Randomized Trial. Pain Res Manag. 2024 Mar 20;2024:9989997. doi: 10.1155/2024/9989997. eCollection 2024. PMID 38550709